CLINICAL TRIAL: NCT02850510
Title: Evaluating a Shortened Version of the Incredible Years Basic Programme in a Non-clinical Community Sample
Brief Title: Evaluating a Shortened Version of the Incredible Years (IY) Basic Programme in a Non-clinical Community Sample
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional centre for children and youth mental health and welfare (Other)
Responsible Party: Principal Investigator, Charlotte Reedtz, Associate professor, Dr. Philos, Regional centre for children and youth mental health and welfare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Shortened version Basic IY
Record Dates: First submitted 2016-07-20; First posted 2016-08-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Parenting Behavior; Child Behavior Problems
Keywords: Harsh discipline; parental competence; positive parenting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief Incredible Years parent training (Experimental): Parent training
  Interventions: Behavioral: Brief Incredible Years parent training
- No parent training (No Intervention): No parent training

INTERVENTIONS:
Behavioral: Brief Incredible Years parent training — The IY parent training programme (3-8 years) developed by Webster-Stratton at the Parenting Clinic, University of Washington, is a manualised and video-based training programme for parents of young children with conduct problems (Webster-Stratton and Reid, 2003a). Parents assigned to the short IY Basic (S-IY) condition were divided into groups of 10-12 parents. The S-IY was led by two experienced group leaders and parents met weekly for two-hour sessions at a public health care center in the community. The group leaders led discussions regarding central aspects of parenting on the basis of the video vignettes, role play and homework.
  Other Names: The Incredible Years Programme series
  Arms: Brief Incredible Years parent training

SUMMARY:
Aim of study:

To evaluate the effects of the shortened version of the Incredible Years (IY) Basic programme, the study which the parents were recruited to. A randomising experimental control between-group design was used with pre- and post-intervention measurements, and a one-year, four-year and ten-year follow-up. Children and families were randomized to either the shortened basic version (n = 89), or the control group (n = 97).

ELIGIBILITY:
Inclusion Criteria:

* No diagnosable behavior problems in child

Exclusion Criteria:

* Diagnosable behavior problems in child

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 189 (Actual)
Dates: Start 2004-01; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Longitudinal change in ECBI scores | baseline, 6-8 weeks after intervention, one-year follow up, four-year follow up, ten-year follow up
  Eyberg Child Behavior Inventory (Robinson et al., 1980). The ECBI provides a list of 36 problem behaviours commonly reported by parents of children with disruptive behaviour problems. The inventory assesses behaviour on two dimensions: the frequency of the behaviour and its identification as a problem. The frequency ratings range from 1 (never) to 7 (always), and are summed to yield an overall problem behaviour Intensity score (Cronbach's alpha 1⁄4 0.82) ranging from 36 to 252.

SECONDARY OUTCOMES:
Reasons for participation and help seeking behaviour | Four-year follow up
  A questionnaire consisting of 12 questions was developed to assess parents' reasons for participating in child rearing classes. Three subscales measure parental concern (five items, a 1⁄4 0.82), motivation to learn (three items, a 1⁄4 0.42), and own/other's opinion (three items, a 1⁄4 0.42). The questionnaire was sent to all participants in the study. Examples of the questions were: ''I was concerned for my child's behaviour'', ''I was uncertain of how to raise my child'', and ''I think it's interesting to learn about children''. All questions were answered using a five-point Likert scale from ''agree'' to ''disagree''.
Longitudinal change in PROC scores | baseline, 6-8 weeks after intervention, one-year follow up, four-year follow up, ten-year follow up
  Parents Sense of Competence (Johnston and Mash, 1989). The PSOC consists of 16 items about parents' confidence on being a parent, answered on a six-point scale ranging from ''strongly disagree'' to ''strongly agree''. Scoring for some items is reversed so that, for all items, higher scores indicate greater parenting self-esteem. Two subscales measure efficacy (seven items, a 1⁄4 0.69) and satisfaction (nine items, a 1⁄4 0.77) in parenting.
Longitudinal change in PSI scores | baseline, 6-8 weeks after intervention, one-year follow up, four-year follow up, ten-year follow up
  Parent Stress Index, Short Form (PSI-SF; Abidin, 1995). The PSI-SF is a 36 item self-report measure of parenting stress, derived from the full version PSI. The PSI-SF yields a total stress (a 1⁄4 0.90) in addition to scores on three scales: parental distress, parent-child dysfunctional interaction, and difficult child.
Longitudinal change in PPI scores | baseline, 6-8 weeks after intervention, one-year follow up, four-year follow up, ten-year follow up
  Parenting Practices Interview (Webster-Stratton et al., 2001). The PPI was adapted from the Oregon Social Learning Centre's Discipline Questionnaire. Two subscales were used; Harsh Discipline (14 items, a 1⁄4 0.79), and Positive Parenting (15 items, a 1⁄4 0.67). Parents reported the probability and the frequency with which they used the different strategies on a seven-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Reedtz, Dr. Philos, Principal Investigator — Arctic University of Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Reedtz C, Klest SK, Aalo NM, Rasmussen ID, Vitterso J. Results From an RCT on Brief Parent Training: Long Term Effects on Parental Quality of Life. Front Psychol. 2019 Feb 18;10:260. doi: 10.3389/fpsyg.2019.00260. eCollection 2019. PMID 30833915
- [Derived] Reedtz C, Klest S. Improved parenting maintained four years following a brief parent training intervention in a non-clinical sample. BMC Psychol. 2016 Aug 24;4(1):43. doi: 10.1186/s40359-016-0150-3. PMID 27553950